CLINICAL TRIAL: NCT01891513
Title: Multimodal Intervention to Reduce Cardiovascular Risk Among Hypertensive Older Adults
Brief Title: ACE Inhibitors Combined With Exercise for Seniors - Pilot Study
Acronym: ACES-P
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500525; 13SDG17080033 (Other Grant/Funding Number: American Heart Association); 099-2013 (Other: Univeristy of Florida)
Record Dates: First submitted 2013-06-24; First posted 2013-07-03 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Hypertension; Aging
Keywords: Physical activity; Hypertension; Physical function; Aging
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Exercise; Angiotensin-Converting Enzyme Inhibitors; Perindopril; Sodium Chloride Symporter Inhibitors; Hydrochlorothiazide; Angiotensin Receptor Antagonists; Losartan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ACE inhibitor + exercise: In addition to exercise training, participants will receive an initial perindopril dose of 4 mg/day which will be titrated to 8 mg/day.
  Interventions: Behavioral: Exercise; Drug: ACE inhibitor + exercise
- Thiazide diuretic + exercise: In addition to exercise training, participants will receive an initial hydrochlorothiazide dose of 12.5 mg/day which will be titrated to 25 mg/day.
  Interventions: Behavioral: Exercise; Drug: Thiazide diuretic + exercise
- Angiotensin receptor blocker + exercise: In addition to exercise training, participants will receive an initial losartan dose of 50 mg/day which will be titrated to 100 mg/day.
  Interventions: Behavioral: Exercise; Drug: Angiotensin receptor blocker + exercise

INTERVENTIONS:
Behavioral: Exercise — All participants will take part in 3 days/week of structured aerobic, stretching, and balance training for weeks 1-12. For weeks, 13-24, training will be reduced to 2 days/week and a resistance training component added. Participants will also be expected to engage in 2 bouts of 30 minutes of home-based walking per week.
Drug: ACE inhibitor + exercise — In addition to exercise training, participants will receive an initial perindopril dose of 2 mg/day which will be titrated to 4 mg/day.
  Other Names: Perindopril
  Groups: ACE inhibitor + exercise
Drug: Thiazide diuretic + exercise — In addition to exercise training, participants will receive an initial hydrochlorothiazide dose of 12.5 mg/day which will be titrated to 25 mg/day.
  Other Names: Hydrochlorothiazide
  Groups: Thiazide diuretic + exercise
Drug: Angiotensin receptor blocker + exercise — In addition to exercise training, participants will receive an initial losartan dose of 50 mg/day which will be titrated to 100 mg/day.
  Other Names: Losartan
  Groups: Angiotensin receptor blocker + exercise

SUMMARY:
The purpose of this study is to compare, when combined with chronic exercise, the effects of perindopril, losartan, and hydrochlorothiazide.

DETAILED DESCRIPTION:
An initial telephone screening will indicate eligibility to participate in the study. The first study visit ("Screening visit") will further determine eligibility to participate. If eligible to fully participate, this study will consist of a structured physical activity program for 24 weeks. In addition, taking daily medication to control your blood pressure and coming to the clinic for several additional assessment visits to monitor your safety and measure study outcomes.

This physical activity program will include moderate-intensity walking, lower-body strengthening, flexibility, and balance training. For the first 12 weeks, of participation there will be three (3) physical activity sessions per week at the physical activity center. These sessions will be led by investigators study staff. These sessions will be used to begin the walking program and to introduce the participant to the strength, stretching, and balance parts of the program in a safe manner. This will allow instructors to better tailor the program to individual needs and abilities. These sessions will involve 40-60 minutes of physical activity instruction. For the final 12 weeks of the intervention, there will be two (2) of these sessions per week.

Participants will also be engage in home-based walking twice per week. This walking can be done at home, community-based physical activity centers (YMCA, senior centers, churches, etc.), or other appropriate facilities as desired. Participants will be asked to report the number of minutes walked each week.

Participants will be randomly assigned to take one of three medications to continue treating blood pressure. These medications are Perindopril, Losartan, and Hydrochlorothiazide. Each medication represents a separate type medication commonly used in practice. These medications are all standard, FDA-approved medications for the treatment of blood pressure. During the time of participating in the study, the use of the normal blood pressure medication will be replaced with the medication assigned during the study. The medications will be inserted into identical capsules by the study pharmacy so that neither participants nor the investigators will know which medication is being used.

Study staff will monitor blood pressure during the study under the supervision of a board-certified cardiologist, and any necessary adjustments to the medication will be indicated by the physician. Participants will also be provided with a blood pressure monitor to use at home during the study and asked to check blood pressure each day and report any abnormal values to study staff. This monitor also automatically records each blood pressure reading. Please bring this monitor to each assessment visit so that study staff can download the stored blood pressure readings.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Hypertension - untreated (Systolic Blood Pressure (SBP) ≥ 140 mm Hg or Diastolic Blood Pressure (DBP) ≥ 90 mm Hg) or treated
* Physical limitations evidenced by either:

Score ≤ 10 on the Short Physical Performance Battery OR Walking speed < 1.2 m/sec during 400 m usual-paced test

* Sedentary lifestyle, defined as <150 min/wk of moderate physical activity as assessed by CHAMPS questionnaire
* Willingness to participate in all study procedures

Exclusion Criteria:

* Failure to provide informed consent
* Inability to complete 400 m walk within 15 minutes without sitting or interpersonal assistance, as an indicator of disablement and likely inability to fully engage in the exercise intervention
* Primary indication for ACE inhibitor use, i.e. Congestive Heart Failure, CAD, diabetes
* Known hypersensitivity to ACE inhibitors
* Resistant hypertension, defined as BP > 140/90, despite the use of three or more anti-hypertensive drugs
* Office or average home SBP > 180 mm Hg or DBP > 110 mm Hg (Average home BP in any seven day period during trial)
* Primary renal disease
* Serum creatinine >2.5 mg/dL in men, or >2.0 mg/dL in women
* Serum potassium >5.0 molar equivalent/L
* Urinary protein > 1 on dipstick
* Abnormal liver enzymes (Aspartate transaminase (AST), Alanine transaminase (ALT), or alkaline phosphatase > 2.5 times the upper limit of normal)
* Severe cardiac disease, including New York Heart Association Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Acute myocardial infarction identified by ECG
* Lives in a nursing home (persons living in assisted or independent housing will not be excluded)
* Significant cognitive impairment, defined as a known diagnosis of dementia or a Mini-Mental State Examination exam score < 24
* Unable to communicate because of severe hearing loss or speech disorder
* Severe visual impairment, which would preclude completion of the assessments and/or intervention
* Other significant co-morbid disease that would prevent participation in exercise
* Planning to move out of the area during the study time frame
* Simultaneous participation in another intervention trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Aging adults with hypertension and physical limitation within Alachua County
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in Walking Speed | Baseline, 6 months
  Investigators will assess walking speed by asking the participants to walk at their usual pace over a 4 m course. Participants will be instructed to stand with both feet touching the starting line and to start walking after a specific verbal command.

SECONDARY OUTCOMES:
Change in body composition | Baseline, 6 months
  Changes in skeletal muscle and adipose tissue (by modulating cardiometabolic function)both fat mass and fat-free mass (FFM) will be assessed using dual energy x-ray absorptiometry (DEXA).
Changes in circulating indices of cardiovascular risk | Baseline, 6 months
  Fasting blood samples (serum or plasma as appropriate) will be evaluated for blood lipids, glucose, and hemoglobin A(1c) levels. Samples will also be used to assay for prominent markers of inflammation (e.g. Tumor necrosis factor-α (TNF-α), Interleukin 6 (IL-6), Vascular cell adhesion protein 1 (VCAM-1), E-selectin) and oxidative stress, including oxidized LDL and myeloperoxidase (MPO).
Change in Exercise Capacity | Baseline, 6 months
  Investigators will assess exercise capacity of participants using the six-minute (6-min) walk test, a safe and reliable test of aerobic endurance in older persons and those with cardiovascular conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Buford, Ph.D., Principal Investigator — University of Florida Department of Aging and Geriatric Research
Locations (1):
- UF Institute on Aging Clinical and Translational Research Building, Gainesville, Florida, United States

REFERENCES:
- See also: University of Florida Institute on Aging — http://aging.ufl.edu